CLINICAL TRIAL: NCT03431610
Title: A Phase 1b Multi-Center, Double-Blind, Randomized Vehicle-Controlled Study Assessing the PK , Pharmacodynamics, Safety and Tolerability of SB414 in Subjects With Atopic Dermatitis
Brief Title: A Phase 1b Study Assessing the PK, PD, Safety & Tolerability of SB414 in Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AD101
Record Dates: First submitted 2018-01-31; First posted 2018-02-13 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SB414 2% (Experimental): SB414 2% topically twice daily
  Interventions: Drug: SB414 2%
- SB414 6% (Experimental): SB414 6% topically twice daily
  Interventions: Drug: SB414 6%
- Vehicle Cream (Placebo Comparator): Vehicle Cream topically twice daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SB414 2% — Twice daily
  Other Names: NVN1000
  Arms: SB414 2%
Drug: SB414 6% — Twice daily
  Other Names: NVN1000
  Arms: SB414 6%
Drug: Vehicle — Placebo comparator
  Other Names: Placebo
  Arms: Vehicle Cream

SUMMARY:
This is a Phase 1b, 2-week study assessing the pharmacokinetics, pharmacodynamics, safety and tolerability of SB414 in subjects with mild to moderate AD.

DETAILED DESCRIPTION:
This is a phase 1b, multi-center, randomized, double-blind, vehicle-controlled study to be conducted in approximately 48 non-immunocompromised adult subjects with mild to moderate AD. Subjects will be randomized to 2 active and 1 vehicle treatment arms. Subjects will apply the study drug (SB414 or Vehicle) to affected areas twice daily for 2 weeks (14 days).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and older, and in good general health;
* EASI score >1 and ≤21, involving ≥5% body surface area (BSA).
* Two target lesions at least 5 cm2 with a TLSS ≥5. Target lesions can not be located on the groin, hands, elbows, feet, ankles, knees, face or scalp.
* Willing to not use any other products for AD during the study;
* Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) prior to randomization and must agree to use an effective method of birth control during the study and for 30 days after their final study visit.

Exclusion Criteria:

* Concurrent or recent use of topical or systemic medications without a sufficient washout period;
* Immunocompromised subjects including those who are known HIV positive or receiving current immunosuppressive treatment,
* Female subjects who are pregnant, nursing mothers, or planning to become pregnant during the study;
* Active acute bacterial, fungal, or viral skin infection within 1 week before the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of hMAP3 | Day 15
  Peak plasma concentrations of hMAP3 after topical application of SB414

SECONDARY OUTCOMES:
Pharmacodynamics of SB414 | Day 15
  Change in relevant Pre and post dose tissue cytokine levels (mg/mg tissue)
Safety Profile (Reported Adverse Events) | Day 15
  Reported Adverse Events
Investigator Assessment of Tolerability | Baseline, Week 1 and Week 2
  Investigator assessment of overall degree of irritation
Subject Assessment of Tolerability | Baseline, Week 1 and Week 2
  Subject-reported from 5 point tolerability scale overall presence and degree of itching and burning / stinging
Efficacy as assessed by EASI (Eczema area and severity index) score | Screening, Baseline and Week 2
  EASI Score will be collected
Efficacy as assessed by Target Lesion Severity Score | Screening, Baseline, Week 1 and Week 2
  Target Lesion Severity Score will be collected
Efficacy as assessed by Itch NRS | Baseline, Week 1 and Week 2
  Itching due to AD as reported by subject on an 11 point numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Maeda-Chubachi, Study Chair — Novan, Inc.
Locations (9):
- United States (9):
  - Novella Site# 242, Coral Gables, Florida
  - Novella Site# 264, Sweetwater, Florida
  - Novella Site# 247, Boise, Idaho
  - Novella Site# 251, Indianapolis, Indiana
  - Novella Site# 201, Berlin, New Jersey
  - Novella Site# 250, Portland, Oregon
  - Novella Site# 265, Hazleton, Pennsylvania
  - Novells Site# 263, Pflugerville, Texas
  - Novella Site# 114, Norfolk, Virginia

REFERENCES:
- [Derived] Guttman-Yassky E, Gallo RL, Pavel AB, Nakatsuji T, Li R, Zhang N, Messersmith E, Maeda-Chubachi T. A Nitric Oxide-Releasing Topical Medication as a Potential Treatment Option for Atopic Dermatitis through Antimicrobial and Anti-Inflammatory Activity. J Invest Dermatol. 2020 Dec;140(12):2531-2535.e2. doi: 10.1016/j.jid.2020.04.013. Epub 2020 May 16. No abstract available. PMID 32428543